CLINICAL TRIAL: NCT05212623
Title: A Single-center, Randomized, Blinded, Positive Controlled Clinical Trial to Assess the Reactogenicity and Immunogenicity of a Quadrivalent Inactivated Influenza Vaccine in Healthy Participants Aged 6-35 Months
Brief Title: A Clinical Trial of an Quadrivalent Inactivated Influenza Vaccine in Healthy Children Aged 6 to 35 Months
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Changchun Institute of Biological Products Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LGYM（SJ）-2021-I
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; quadrivalent influenza split vaccine; reactogenicity; immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Subjects received 2 doses of 0.25 mL of quadrivalent influenza vaccine, 4 weeks apart.
  Each 0.25-ml dose contained 7.5 μg of hemagglutinin per strain (Four types of virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata).
  Interventions: Biological: quadrivalent influenza split vaccine
- Group B (Experimental): Subjects received 2 doses of 0.5 mL of quadrivalent influenza vaccine, 4 weeks apart. Each 0.5-ml dose contained 15 μg of hemagglutinin per strain.(Four types of virus strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata).
  Interventions: Biological: quadrivalent influenza split vaccine
- Group C (Active Comparator): Subjects received 2 doses of 0.25 mL of influenza vaccine, 4 weeks apart. Each 0.25-ml dose contained 7.5 μg of hemagglutinin per strain (3 type of virus strains, including BY).
  Interventions: Biological: Influenza virus split vaccine
- Group D (Active Comparator): Subjects received 2 doses of 0.25 mL of influenza vaccine, 4 weeks apart. Each 0.25-ml dose contained 7.5 μg of hemagglutinin per strain (3 types of virus strains, including BV).
  Interventions: Biological: Influenza virus split vaccine

INTERVENTIONS:
Biological: quadrivalent influenza split vaccine — This vaccine is produced by Changchun Sponsor Institute of Biological Products Co., Ltd. Subjects will receive two doses of quadrivalent influenza vaccine administered 4 weeks apart by intramuscular injection
  Arms: Group A
Biological: quadrivalent influenza split vaccine — This vaccine is produced by Changchun Sponsor Institute of Biological Products Co., Ltd. Subjects will receive two doses of quadrivalent influenza vaccine administered 4 weeks apart by intramuscular injection
  Arms: Group B
Biological: Influenza virus split vaccine — This vaccine is produced by Changchun Sponsor Institute of Biological Products Co., Ltd. Subjects will receive two doses of quadrivalent influenza vaccine administered 4 weeks apart by intramuscular injection
  Arms: Group C
Biological: Influenza virus split vaccine — This vaccine is produced by Changchun Sponsor Institute of Biological Products Co., Ltd. Subjects will receive two doses of quadrivalent influenza vaccine administered 4 weeks apart by intramuscular injection.
  Arms: Group D

SUMMARY:
In this single-center, randomized, blinded, positive-controlled design, the investigators will assess the safety and immunogenicity of 2 doses of an inactivated quadrivalent influenza vaccine in children aged 6 to 35 months.

About 120 healthy participants are planned to be enrolled, of who 60 participants were enrolled in the low-dose group and 60 participants were enrolled in the high-dose group. In the low-dose group, participants were randomly (2:1:1) assigned to receive a quadrivalent inactivated influenza vaccine (IIV4) at 0.25 mL including A/H1N1, A/H3N2, B/Victoria, and B/Yamagata, and a trivalent inactivated influenza vaccine (IIV3) at 0.25 mL including A/H1N1, A/H3N2 and B/Victoria, and IIV3 at 0.25 mL including A/H1N1, A/H3N2, and B/Yamagata. In the high-dose group, participants were randomly (2:1:1) assigned to receive IIV4 at 0.5 mL, and IIV3 at 0.25 mL including A/H1N1, A/H3N2, and B/Victoria, and IV3 at 0.25 mL including A/H1N1, A/H3N2, and B/Yamagata. Subjects receive 2 doses of influenza vaccine 4 weeks apart.

The occurrence of adverse reactions within 30 minutes, the occurrence of adverse reactions within 28 days, and serious adverse events within 6 months after vaccination will be observed in all participants. For participants aged 24-35 months in each dose group, laboratory safety tests were measured before enrollment and on day 4 post each dose to assess any toxic effects. In addition, all subjects will be required to collect blood for HI antibody testing before the first dose of vaccination and 30 days after the second dose of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants and young children aged 6-35 months, provide vaccination certificate and birth medical certificate.
* The subject or legal guardian can provide with informed consent and sign the informed consent form.
* The subjects or legal guardians are able to and willing to use a thermometer, a scale and fill in a diary card/contact card as required, and be able to comply with the requirements of the clinical trial protocol to complete clinical research.

Exclusion Criteria:

1. st dose:

   * Axillary temperature>37.0℃
   * Participants aged 24-35 months, with abnormal blood routine, blood biochemical and urine routine indexes and judged by the researchers as having clinical significance.
   * Influenza within the past 3 months (confirmed clinically, serologically or microbiological).
   * Have previously received any influenza vaccine (registered or experimental) or planned to receive any influenza vaccine during the study.
   * Allergy to any component of the study vaccine, history of allergic reaction to eating eggs or using gentamicin sulfate.
   * History of severe allergies to any vaccines or drugs.
   * Preterm (delivered before 37 weeks of gestation), low birth weight (birth weight <2500g) infants (only for volunteers aged 6 months to 12 months).
   * Dystocia, suffocation rescue, nervous system damage history.
   * Congenital malformations or developmental disorders affecting organ function, genetic defects, severe malnutrition, etc..
   * Acute illness, severe chronic illness, or acute exacerbation of chronic illness on the day of vaccination.
   * History of vaccination with the live attenuated vaccine within 14 days prior to vaccination and other vaccination within 7 days.
   * Those receiving immune enhancement or inhibitor therapy within 3 months (continuous oral or infusion for more than 14 days).
   * Have congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases.
   * History of asthma, unstable in the past two years requiring urgent treatment, hospitalization, intubation, oral or intravenous corticosteroids.
   * Receive blood or blood-related products within 3 months.
   * Have a medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
   * History of coagulation abnormalities (eg, coagulation factor deficiency, coagulation disorder)
   * Plan to relocate before the end of the study or to be away from home for an extended period of time during scheduled study visits
   * Participating in or planning to participate in other clinical trials in the near future
   * Abnormal laboratory test indicators, except for minor abnormalities that have no clinical significance as judged by the doctor.
   * The investigator judges any situation that is inappropriate to participate in this clinical trial
2. nd dose:

   * Severe allergic reaction after the first dose of the vaccine.
   * Serious adverse reactions causally related to the first dose of the vaccine.
   * After the first vaccination, newly discovered or newly occurred do not meet the first-dose inclusion criteria or meet the first-dose exclusion criteria will be determined by the investigator whether to continue participating in the study.
   * Other reasons for exclusion in the opinion of the investigator.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events within 7 days after each vaccination in the participants aged 6-35 months. (Including abnormal laboratory test indicators and clinical significance) | On day 7 after each dose
  Incidence of adverse events within 7 days after each vaccination in the participants aged 6-35 months. (Including abnormal laboratory test indicators and clinical significance)

SECONDARY OUTCOMES:
Incidence of adverse events from the first dose to 30 days after the second dose in the participants aged 6-35 months. | Time Frame: within 30 days after the second dose
  Incidence of adverse events from the first dose to 30 days after the second dose in the participants aged 6-35 months.
Incidence of serious adverse events (SAE) till the 6 months after the second dose in the participants aged 6-35 months. | within 6 months after the second dose
  Incidence of serious adverse events (SAE) till the 6 months after the second dose in the participants aged 6-35 months.
HI antibody-positive conversion rate in each group 30 days after the second vaccination in the participants aged 6-35 months. | on day 30 after the second vaccination
  HI antibody-positive conversion rate in each group 30 days after the second vaccination in the participants aged 6-35 months.
Seroprotection rate 30 days after the second dose in each group in the participants aged 6-35 months. | on day 30 after the second vaccination
  Seroprotection rate 30 days after the second dose in each group in the participants aged 6-35 months.
GMT of HI antibodies 30 days after the second dose of each group in the participants aged 6-35 months. | on day 30 after the second vaccination
  GMT of HI antibodies 30 days after the second dose of each group in the participants aged 6-35 months.
GMI of HI antibodies 30 days after the second dose of each group in the participants aged 6-35 months. | on day 30 after the second vaccination
  GMI of HI antibodies 30 days after the second dose of each group in the participants aged 6-35 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Centers for Disease Control and Prevention, Nanjing, Jiangsu, China